CLINICAL TRIAL: NCT00017992
Title: An Open-Label Study of a Once Daily Dose of Emtricitabine in Combination With Other Antiretroviral Agents in HIV-Infected Pediatric Patients
Brief Title: Emtricitabine Given Once A Day With Other Anti-HIV Drugs in Children With HIV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Triangle Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 298D; FTC-203
Record Dates: First submitted 2001-06-23; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Administration Schedule; Stavudine; HIV Protease Inhibitors; Ritonavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; ABT 378; emtricitabine
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Emtricitabine; Stavudine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Emtricitabine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if emtricitabine is safe in children infected with HIV and to determine the best dose.

DETAILED DESCRIPTION:
Children are placed into 1 of 4 treatment groups based on age: Group 1, 3 months to 24 months; Group 2, 25 months to 6 years; Group 3, 7 years to 12 years; Group 4, 13 years to 17 years. They receive baseline evaluations. Antiretroviral-naive patients receive emtricitabine plus stavudine plus lopinavir/ritonavir. Antiretroviral-experienced patients replace lamivudine with emtricitabine. Patients return to the clinic for follow-up visits at Weeks 2 and 4 and then every 4 weeks until Week 48. Safety is evaluated using adverse events, which are reviewed at every clinic visit. Clinical laboratory data and full-profile pharmacokinetics of emtricitabine are evaluated at some visits. After the Week 48 study evaluations are completed, individual patients may continue to receive study medication (as provided by the sponsor) until commercially available, if certain criteria are met.

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are at least 3 months old and no older than 17 years of age. This is the age the child needs to be at the time they begin the study.
* Are HIV positive.
* Weigh more than 5.5 pounds. A newborn child must have reached at least 38 weeks of gestation.
* Have or have not taken anti-HIV drugs. Those that have not must have a viral load between 5,000 and 500,000 copies/ml at screening. Those that have must have been taking anti-HIV drugs, including lamivudine, for at least 3 months and have a viral load of no more than 400 copies/ml at screening.
* Have a CD4 count of more than 200 cells/mm3.
* Have written consent from parent or guardian.
* Are willing to use effective birth control during the study and for 1 month after the last dose of emtricitabine, if sexually active.

Exclusion Criteria

Children will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Cannot follow the visit or dosing schedule or are not available for 1 year.
* Have taken experimental drugs or vaccines (except for emivirine and experimental forms of approved drugs) within 30 days of study start.
* Have nerve damage in their arms or legs.
* Have trouble eating or taking drugs.
* Have serious diarrhea within 30 days before study entry.
* Have had any serious illness within 30 days of study screening. Any treatment must have been finished 14 days before study entry.
* Have had an AIDS-related (opportunistic) disease within 12 months of screening.
* Are being treated for tuberculosis.
* Have had pancreatitis.
* Require certain drugs.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100

CONTACTS AND LOCATIONS:
Locations (14):
- United States (8):
  - USC School of Medicine / LA County Med Ctr, Los Angeles, California
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami, Miami, Florida
  - New York Hosp / Cornell Med Ctr, New York, New York
  - St Luke's - Roosevelt Hosp Ctr, New York, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
- Fundacion HUES, Buenos Aires, Argentina
- Instituto Mexicano de Investigacion Clinica, Colonia Roma, Mexico
- Hospital del Nino, Panama City, Panama
- Univ of Puerto Rico / Med Science Campus, San Juan, Puerto Rico
- South Africa (2):
  - Perinatal HIV Research UNIT, Diepkloof
  - Infectious Diseases Clinincal Trial Unit, Gaunteng